CLINICAL TRIAL: NCT06788548
Title: Fluorescence Guided Laparoscopic-Endoscopic Cooperative Sentinel Lymph Node Navigation Surgery Strategy for Early Gastric Cancer: A Multicenter Randomized Controlled Trial Study
Brief Title: Fluorescence Guided Laparoscopic-Endoscopic Cooperative Sentinel Lymph Node Navigation Surgery Strategy for Early Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: China-Japan Friendship Hospital (Other); Cancer Hospital Chinese Academy of Medical Scienc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRWEP2024W162020112; 7232334 (Other Grant/Funding Number: Beijing Natural Science Foundation); D171100006517003 (Other Grant/Funding Number: Beijing Municipal Science & Technology Commission); PX2020001 (Other Grant/Funding Number: Beijing Municipal Administration of Hospitals Incubating Program); PX20240103 (Other Grant/Funding Number: Beijing Municipal Administration of Hospitals Incubating Program); No.2024-2-2028 (Other Grant/Funding Number: Capital's Funds for Health Improvement and Research); Z241100007724004 (Other Grant/Funding Number: Beijing Municipal Science & Technology Commission AI+ Health Collaborative Innovation Cultivation Project); BRWEP2024W162020100 (Other Grant/Funding Number: Beijing Research Ward Excellence Program, BRWEP); BRWEP2024W162020112 (Other Grant/Funding Number: Beijing Research Ward Excellence Program, BRWEP); YC202401QX0824 (Other Grant/Funding Number: Excellent Plan for Medicine Innovation and Translation project); 82300646 (Other Grant/Funding Number: National Natural Science Foundation of China); [ZHKY-2025-1869（B012）] (Other Grant/Funding Number: Beijing Integrated Medical Association Clinical Research Funding Program); No.2024ZD0520600 (Other Grant/Funding Number: Noncommunicable Chronic Diseases-National Science and Technology Major Project Award)
Record Dates: First submitted 2024-12-16; First posted 2025-01-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-01

CONDITIONS: Early Gastric Cancer
Keywords: Early Gastric Cancer; Sentinel Lymph Node; Basin Dissection; Laparoscopic surgery; Safety AND Efficacy; Fluorescence Guided; Laparoscopic-Endoscopic Cooperative Surgery; multicenter
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluorescence Guided Laparoscopic-Endoscopic Cooperative Sentinel Lymph Node Navigation Surgery Strat (Experimental): Laparoscopic-endoscopic cooperative surgery (LECS) offers a more targeted approach through the integration of the complementary strengths of endoscopy and laparoscopy. LECS enables accurate targeting, optimal resection margins and tissue sparing excision. Consequently, LECS better preserves gastric architecture and function, potentially leading to enhanced postoperative recovery and QoL. Nevertheless, current evidence supporting LECS for SNNS remains limited.
  Interventions: Procedure: Fluorescence Guided Laparoscopic-Endoscopic Cooperative Sentinel Lymph Node Navigation Surgery
- D2 gastrectomy (Active Comparator): A preoperative contrast-enhanced abdominal CT scan is conducted to assess the lesion's location, tumor dimensions, and lymph node metastasis (LNM). Preoperative endoscopic dye injection or intraoperative endoscopic localization is utilized to accurately identify the tumor site and ensure adequate resection margins. The extent of lymph node dissection (LND) adheres to the Japanese gastric cancer treatment guidelines 2023 (6th edition)[4]. Specifically, D2 distal gastrectomy encompasses lymph nodes No. 1, 3, 4sb, 4d, 5, 6, 7, 8a, 9, 11p, and 12a. D2 proximal gastrectomy includes nodes 1, 2, 3a, 4sa, 4sb, 7, 8a, 9, 11p, and 12a, while D2 total gastrectomy involves nodes 1, 2, 3, 4sa, 4sb, 4d, 5, 6, 7, 8a, 9, 11p, 11d, and 12a.
  Interventions: Procedure: Laparoscopic D2 radical gastrectomy

INTERVENTIONS:
Procedure: Fluorescence Guided Laparoscopic-Endoscopic Cooperative Sentinel Lymph Node Navigation Surgery — Patients without prior ESD received ESD with laparoscopic sentinel basin dissection (LSBD) for ESD resectable lesions, otherwise patients received laparoscopic-endoscopic cooperative regional gastrectomy (LRG) with LSBD. For patients with prior non-curative ESD, LSBD alone was performed if margins were negative, otherwise LRG with LSBD was conducted.
  LECS-SNNS adopted a left-sided surgical approach. During laparoscopic sentinel node basin dissection (LSBD), indocyanine green (ICG) (2 mL, 2.5 mg/mL) was endoscopically injected into the submucosal layer at four quadrants around the marking points (0.5 mL per quadrant). Sentinel lymph node basins (SLBs) were defined as the area within a 2 cm margin of the detected fluorescence stained nodes, which were marked with laparoscopic clips.
  Fifteen minutes after ICG injection, the SLBs were examined first under white light and then using fluorescence imaging. Staining status was determined by consensus among surgeons and endoscopists.
  Arms: Fluorescence Guided Laparoscopic-Endoscopic Cooperative Sentinel Lymph Node Navigation Surgery Strat
Procedure: Laparoscopic D2 radical gastrectomy — Preparation: The patient is positioned supine with general anesthesia. An orogastric tube and Foley catheter are inserted. Antibiotics are administered, and sequential stockings are applied. Port Placement: Pneumoperitoneum is created via a Veress needle at the umbilicus. Working ports are placed in the upper quadrants, with a fifth port for liver retraction. Abdominal Exploration: The abdomen is inspected for metastases, and peritoneal cytology is performed. Dissection and Lymph Node Removal: The lesser omentum is divided near the liver, reaching the cardia and diaphragm. The gastrocolic ligament is divided along the transverse colon. Lymph node dissection begins along the splenic artery, then proceeds to the left gastric artery and celiac nodes. The left gastric vessels are controlled with endoclips.After lymph node dissection, distal subtotal gastrectomy is performed. Digestive tract reconstruction is typically done through a mini-laparotomy.
  Arms: D2 gastrectomy

SUMMARY:
The main treatment for early gastric cancer (EGC) include endoscopic submucosal dissection (ESD) and radical gastrectomy. However, appropriate treatment for patients who exceed the absolute indications and noncurative resection of ESD remains unestablished. Sentinel node navigation surgery (SNNS) enables limited lymph node resection, thereby facilitating function-preserving gastrectomy (FPG) and improving quality of life (QoL). SNNS seems to be the promising solution according to previous study, however evidence-based medicine was lacking. It is imperative to establish its safety and efficacy in patients with EGC. However, the optimal implementation of FPG remain unclear. Moreover, objective assessment of postoperative functional outcomes,remains limited.

DETAILED DESCRIPTION:
The main treatment for early gastric cancer (EGC) include endoscopic submucosal dissection (ESD) and radical gastrectomy. However, appropriate treatment for patients who exceed the absolute indications and noncurative resection of ESD remains unestablished. Sentinel node navigation surgery (SNNS) enables limited lymph node resection, thereby facilitating function-preserving gastrectomy (FPG) and improving quality of life (QoL). SNNS seems to be the promising solution according to previous study, however evidence-based medicine was lacking. It is imperative to establish its safety and efficacy in patients with EGC. However, the optimal implementation of FPG remain unclear. Moreover, objective assessment of postoperative functional outcomes,remains limited.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients aged 18-80 years, regardless of gender. 2) Patients with Eastern Cooperative Oncology Group (ECOG) score ≤ 2 and American Society of Anesthesiologists (ASA) score ≤ 2 who are candidates for a curative D2 gastrectomy.

  3) Patients without prior gastrointestinal surgery, chemotherapy, or radiotherapy.

  4) Patients with normal liver, kidney, heart, lung, and bone marrow function (GPT × 109 /L, PLT>109 /L).

  5) Patients capable of understanding and adhering to the research protocol. 6) Patients who can provide written informed consent, either personally or through legal representative.

  7) Patients with cT1N0M0 gastric cancer or after non-curative ESD resection, according to the UICC TNM staging system, 8th edition.

Exclusion Criteria:

* 1) Patients with a contraindication for gastroscopy. 2) Patients with uncontrollable diseases, such as coagulation disorders, epilepsy, central nervous system diseases or mental disorders, cardiopulmonary insufficiency, unstable angina, myocardial infarction, a cerebrovascular accident that occurred within 6 months, and other surgical contraindications.

  3) Patients unable to undergo general anesthesia or surgical treatment due to conditions related to other organs, or unwilling to undergo surgery.

  4) Patients with gastric stump cancer, recurrent gastric cancer, multiple primary malignant tumors in the abdominopelvic cavity, or a history of other malignant tumors within the previous 5 years.

  5) Pregnant or lactating women. 6) Participants enrolled in other clinical trials. 7) Patients with undeterminable tracer staining range or contraindications to tracer use.

  8) Patients who fail to receive or fail ESD therapy. 9) Patients who meet the absolute indication of ESD.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
3 and 5-year disease free survival | From treatment to 3 and 5-years after surgery

SECONDARY OUTCOMES:
5-year overall survival | From treatment to 5-years after surgery
Mortality (within 30 days after surgery)；Unscheduled second surgery (within 30 days after surgery) and Unplanned return to hospital (within 30 days after surgery) | From treatment to 30-days after surgery
rate of inconsistent result between intraoperative rapid pathology and postoperative pathology examine；Rates of remedial and additional surgery | From enrollment to 1 week after surgery
Perioperative complication rate (within 30 days after surgery, including bleeding, perforation, lymphatic leakage, respiratory complications, cardiovascular complications, anastomotic fistula | From treatment to 30-days after surgery
  According to the Clavien-Dindo scale, if the postoperative complication grade is higher than grade II, it is considered clinically significant)
Operation time | From treatment to 1 week after surgery
R0 resection rate | From treatment to 1 week after surgery
additional surgical operation rate | From treatment to 5-years after surgery
blood loss | From treatment to 30-days after surgery
postoperative length of stay | From treatment to 30-days after surgery
overall hospitalization cost | From treatment to 5-years after surgery
Gastric emptying scintigraphy result | From treatment to 5-years after surgery
date of gas evacuation | From treatment to 30-days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No